CLINICAL TRIAL: NCT06209476
Title: Clinical Investigation on Assessing the Repeatability and Reproducibility of Central and Peripheral Refractive Error Measurement With the Grand Seiko WAM-5500
Brief Title: Clinical Investigation on Assessing the Repeatability and Reproducibility of Central and Peripheral Refractive Error
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6559
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Experimental — Eligible subjects with sphere component of the subjective spherocylindrical refraction between +1.50 to -6.00D (inclusive) and 2.00D or less astigmatism in the right eye will be unilaterally measured with the WAM-5500 autorefractor by 3 testers.

SUMMARY:
This is a unilateral, non-interventional study. Each subject will be unilaterally measured with the WAM-5500 autorefractor by 3 testers. All measurements will be made on the right eye only.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 50 (inclusive) years of age at the time of screening.
4. The spherical component of the subject's non-vertex-corrected distance subjective refraction must be between +1.50 and -6.00DS (inclusive), with the magnitude of the cylinder 2.00 DC or less in the right eye.
5. The subject must have a Van Herrick angle grade of at least 3 or greater in the right eye.
6. The subject must have a BSCVA of at least 20/30 (defined as reading at least 3 out of the 5 letters on the 20/30 line) in the right eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be diabetic or pre-diabetic by self-report.
3. Have a history of ocular trauma, systemic disease or medication use known to cause variability in refractive error.
4. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, scleral lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 3 months.
6. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
7. Take ocular and systemic medications known to interact with Tropicamide ophthalmic solution or systemic medications that can cause myopia.
8. Have a history of an allergic reaction to Tropicamide or Proparacaine.
9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities, or bulbar injection) or other corneal or ocular disease or abnormalities that may compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, corneal scar or opacity ≥ 0.3 mm, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
10. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
11. Have a history of strabismus, amblyopia, nystagmus, or any condition that affects fixation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female subjects between 18 and 50 years of age (inclusive) of any ethnicity with sphere component of the subjective spherocylindrical refraction between +1.50 to -6.00D (inclusive) and 2.00D or less astigmatism in the right eye.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Central (on-axis) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Central (on-axis) cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of central refractive error measurements with the Grand Seiko WAM-5500.
Peripheral (10° off-axis on the temporal retina) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 10° temporal retina.
Peripheral (20° off-axis on the temporal retina) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 20° temporal retina.
Peripheral (30° off-axis on the temporal retina) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 30° temporal retina.
Peripheral (10° off-axis on the nasal retina) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 10° nasal retina.
Peripheral (20° off-axis on the nasal retina) cycloplegic auto-refraction: | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 20° nasal retina.
Peripheral (30° off-axis on the nasal retina) cycloplegic auto-refraction | Up to 10-day follow-up visit
  Peripheral cycloplegic auto-refraction will be measured to evaluate the intra-visit repeatability, inter-visit repeatability, and reproducibility of peripheral refractive error measurements with the Grand Seiko WAM-5500 at 30° nasal retina.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- VRC, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu